CLINICAL TRIAL: NCT05838157
Title: Research for the Effect of HPV Vaccine on Menstrual Cycle in Women of Reproductive Age
Brief Title: The Effect of HPV Vaccine on Menstrual Cycle in Women of Reproductive Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao Juan, Attending physician, Sun Yat-sen University
Other Study IDs: 2022111615154477
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Menstrual Disorder; Premature Ovarian Failure
Keywords: HPV vaccine; menstrual cycle; menstrual disorder; premature ovarian insufficiency
MeSH Terms: conditions — Menstruation Disturbances; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Girls and women aged 16 to 40 years who receiving at least one dose of HPV vaccination: Girls and women aged 16 to 40 years who receiving HPV vaccination ( including 2vHPV、4vHPV、9vHPV) in Cancer Prevention Center, Sun Yat-sen University Cancer Center during April 10th 2023 to April 30th 2023.
  Interventions: Biological: prophylactic HPV vaccine(bivalent HPV、quadrivalent HPV、9-valent HPV)

INTERVENTIONS:
Biological: prophylactic HPV vaccine(bivalent HPV、quadrivalent HPV、9-valent HPV) — at least one dose of prophylactic HPV vaccine including bivalent HPV (2vHPV)， quadrivalent HPV vaccine (4vHPV)，9-valent HPV vaccine (9vHPV)

SUMMARY:
Cervical cancer is one of the most common cancer in women, making it the fourth largest cause of female cancer mortality worldwide. High-risk HPV types (hrHPV) continuous infection is the main cause of the premalignant and malignant lesions of the cervix. The most effective primary prevention of cervical cancer is administration HPV vaccines. There are three prophylactic HPV vaccines including bivalent HPV (2vHPV)， quadrivalent HPV vaccine (4vHPV)，9-valent HPV vaccine (9vHPV) currently. With the widespread of HPV vaccination， the cases related to abnormal menstrual cycle or menstrual irregularities has gradually increased in the Vaccine Adverse Event Reporting System, also the number of reports and studies were increasing. We designed this study to evaluate the statistical association of HPV vaccine and changes in menstrual cycle or menstrual irregularities、amenorrhea. And detect the signal of premature ovarian insufficiency (POI) and related events of three HPV vaccines, and to provide evidence for the safety of HPV vaccines based on the data mining and signal detection method. The research data was obtained from prospective self- developed questionnaire. Before-after study was applied in this study, investigators collect the menstrual cycle data of subjects by the questionnaire and qualitatively interview were taken. The control group is before vaccination, HPV vaccination is Intervention group.

DETAILED DESCRIPTION:
High-risk HPV types (hrHPV) continuous infection is the main cause of the premalignant and malignant lesions of the cervix. The most effective primary prevention of cervical cancer is administration HPV vaccines. There are three prophylactic HPV vaccines including bivalent HPV (2vHPV)， quadrivalent HPV vaccine (4vHPV)，9-valent HPV vaccine (9vHPV) currently. With the widespread of HPV vaccination， the cases related to abnormal menstrual cycle or menstrual irregularities has gradually increased in the Vaccine Adverse Event Reporting System, also the number of reports and studies were increasing. Whereas all of the studies are retrospective and the data from passive surveillance system, meanwhile, HPV vaccines has been available in Chinese mainland less than 7 years. Especially, 9vHPV applicable range was broadened to 45 years shortly before. There are rarely prospective researches focus on the connection between HPV vaccines and menstrual disorder. We designed this prospective study to observe and evaluate the statistical association of HPV vaccine and menstrual disorder such as menstrual irregularities、amenorrhea、 hypomenorrhea or hypermenorrhea in Chinese women. And detect the signal of premature ovarian insufficiency (POI) and related events of three HPV vaccines, and to provide evidence for the safety of HPV vaccines based on the data mining and signal detection method.

The study design used self-control, We using a self-designed questionnaire collect the menstruation data of girls and women aged 16 to 40 years who receiving HPV vaccination ( including 2vHPV、4vHPV、9vHPV) in Cancer Prevention Center, Sun Yat-sen University Cancer Center during May 10th 2023 to April 30th 2023. The self-designed questionnaire contains three parts. First part includes personal basic information such as age, profession, education Level, marital or childbearing status etc. Part two there are containing health status, menstruation conditions (include menstrual cycle, menstrual period, menstrual blood volume and dysmenorrhea etc). Part three collects menstruation conditions by qualitatively interview , covers each menstrual cycle after the first dose of HPV vaccination until 3 months after the third dose .

To analyze the data, R studio statistical software was used. The general measurement data were analyzed by paired sample T test, p=0.05. Bayesian trusted Propagation neural network (BCPNN) and multi-item gamma Poisson contractor (MGPS) were used to detect the signals of POI related events and to conduct empirical Bayes data mining among ours database.

ELIGIBILITY:
Inclusion Criteria:

* Previous menstrual cycles were regular and normal
* At least one vaccination of HPV vaccine

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Record of abnormal results of HPV test/ cervical cytology/ gynecological ultrasonography
* Record of medications related to menstruation
* Diseases contribute to menstrual irregularities、amenorrhea such as severe anemia/ coagulation disorders/ thyroid dysfunction etc.
* Participation in other clinical trials

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Girls and women aged 16 to 40 years who receiving HPV vaccination ( including 2vHPV、4vHPV、9vHPV) in Cancer Prevention Center, Sun Yat-sen University Cancer Center during April 10th 2023 to April 30th 2023.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of the menstrual cycle | 3 months after the administration of the third dose of vaccine( starts with the first dose of HPVvaccine, no less than 9 cycles)
  In 16~40 years old women , any frequency shorter than 21 days or longer than 36 days will be defined as abnormal
Duration of the menstrual cycle | 3 months after the administration of the third dose of vaccine( starts with the first dose of HPVvaccine, no less than 9 cycles)
  In 16~40 years old women , any duration shorter than 3 days or longer than 7 days will be defined as abnormal
Quantity of the menstrual cycle | 3 months after the administration of the third dose of vaccine( starts with the first dose of HPVvaccine, no less than 9 cycles)
  In 16~40 years old women , any quantity less than 30 ml or more than 80 ml will be defined as abnormal

SECONDARY OUTCOMES:
Premature ovarian failure (POF) signals | 3 months after the administration of the third dose of vaccine( starts with the first dose of HPVvaccine, no less than 9 cycles)
  From the first dose of the vaccine, Blood biochemical detection used to measure the levels of follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), progesterone (P), testosterone (T) and prolactin (PRL). And Ultrasonography is used to detected changes in the endometrium after each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Xiao, Master, Study Director — Sun Yat-sen University; Chuanbo Xie, PhD, Study Director — Sun Yat-sen University; Junjie Chen, Bachelor, Principal Investigator — Sun Yat-sen University; Huiping Ye, Bachelor, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Cancer Prevention Center,Sun Yat-sen University Cancer Cente, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Cente, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] de Sanjose S, Delany-Moretlwe S. HPV vaccines can be the hallmark of cancer prevention. Lancet. 2019 Aug 10;394(10197):450-451. doi: 10.1016/S0140-6736(19)30549-5. Epub 2019 Jun 26. No abstract available. PMID 31255298
- [Result] Gong L, Ji HH, Tang XW, Pan LY, Chen X, Jia YT. Human papillomavirus vaccine-associated premature ovarian insufficiency and related adverse events: data mining of Vaccine Adverse Event Reporting System. Sci Rep. 2020 Jul 1;10(1):10762. doi: 10.1038/s41598-020-67668-1. PMID 32612121
- [Result] Hviid A, Myrup Thiesson E. Association Between Human Papillomavirus Vaccination and Primary Ovarian Insufficiency in a Nationwide Cohort. JAMA Netw Open. 2021 Aug 2;4(8):e2120391. doi: 10.1001/jamanetworkopen.2021.20391. PMID 34436612
- [Result] Colafrancesco S, Perricone C, Tomljenovic L, Shoenfeld Y. Human papilloma virus vaccine and primary ovarian failure: another facet of the autoimmune/inflammatory syndrome induced by adjuvants. Am J Reprod Immunol. 2013 Oct;70(4):309-16. doi: 10.1111/aji.12151. Epub 2013 Jul 31. PMID 23902317
- [Result] Tatang C, Arredondo Bisono T, Bergamasco A, Salvo F, Costa Clemens SA, Moride Y. Human Papillomavirus Vaccination and Premature Ovarian Failure: A Disproportionality Analysis Using the Vaccine Adverse Event Reporting System. Drugs Real World Outcomes. 2022 Mar;9(1):79-90. doi: 10.1007/s40801-021-00271-6. Epub 2021 Sep 12. PMID 34510402
- [Result] Torella M, Marrapodi MM, Ronsini C, Ruffolo AF, Braga A, Frigerio M, Amabile E, Vastarella MG, Rossi F, Riemma G. Risk of Premature Ovarian Insufficiency after Human Papilloma Virus Vaccination: A PRISMA Systematic Review and Meta-Analysis of Current Evidence. Vaccines (Basel). 2023 Jan 9;11(1):140. doi: 10.3390/vaccines11010140. PMID 36679985
- [Result] Little DT, Ward HR. Adolescent Premature Ovarian Insufficiency Following Human Papillomavirus Vaccination: A Case Series Seen in General Practice. J Investig Med High Impact Case Rep. 2014 Oct 28;2(4):2324709614556129. doi: 10.1177/2324709614556129. eCollection 2014 Oct-Dec. PMID 26425627